CLINICAL TRIAL: NCT02607709
Title: Lymphadenectomy in Urothelial Carcinoma in the Renal Pelvis and Ureter
Brief Title: Lymphadenectomy in Urothelial Carcinoma
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusions
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Urologist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG-79-2015
Record Dates: First submitted 2015-11-15; First posted 2015-11-18 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Ureteral Neoplasms
MeSH Terms: conditions — Ureteral Neoplasms | interventions — Lymph Node Excision; Nephroureterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nephroureterektomy (Placebo Comparator): scheduled to receive routine standard open or robot assisted nephroureterectomy without lymphadenectomy
  Interventions: Procedure: Nephroureterectomy without lymphadenectomy
- Nephroureterektomy + Lymphadenectomy (Experimental): scheduled to received mapped lymphadenectomy in conjugation with nephroureterectomy
  Interventions: Procedure: Lymphadenectomy in conjugation with nephroureterectomy

INTERVENTIONS:
Procedure: Lymphadenectomy in conjugation with nephroureterectomy — Lymphadenectomy (intervention group only):
  Lymphadenectomy performs in four fractions on the right side and two fractions on the left side according to Dissection template (Appendix 1). Renal hilar nodes are included in fraction 1 and 3, respectively.
  Arms: Nephroureterektomy + Lymphadenectomy
Procedure: Nephroureterectomy without lymphadenectomy — Removing the kidney, ureter and bladder cuff
  Arms: Nephroureterektomy

SUMMARY:
Two out of three tumours in the upper urinary tract are located in the renal pelvis. Muscle-invasive urothelial carcinoma is probably more common among tumours in the upper urinary tract compared to tumours in the urinary bladder. Thus, muscle-invasive tumours represent approximately 45 % of renal pelvic tumours compared to 25 % of tumours within the urinary bladder. As in the bladder, lymph node metastases are rare in non-muscle invasive disease. Information regarding indications, extent and possible curative potential is currently lacking for lymphadenectomy in conjunction with nephroureterectomy for urothelial carcinoma in the upper urinary tract (UUTUC). There are, however, retrospective series with survival data for patients with lymph node metastasis that report long term survival after surgery as monotherapy [4] with similar survival proportions as in bladder cancer with lymph node metastases after radical cystectomy. A retrospective study from Tokyo was expanded to the only available prospective study, where 68 patients with UUTUC were submitted to template-based lymphadenectomy. Another retrospective study by the same Japanese group, showed that 5-year cancer-specific and recurrence-free survival was significantly higher in the complete lymphadenectomy group than in the incomplete lymphadenectomy or without lymphadenectomy groups. Tanaka N et al. reported recurrence rate after nephroureterectomy without lymphadenectomy at 1 and 3 years were 18.9 and 29.8 %, respectively.

DETAILED DESCRIPTION:
Background:

Two out of three tumours in the upper urinary tract are located in the renal pelvis. Muscle-invasive urothelial carcinoma is probably more common among tumours in the upper urinary tract compared to tumours in the urinary bladder. Thus, muscle-invasive tumours represent approximately 45 % of renal pelvic tumours compared to 25 % of tumours within the urinary bladder. As in the bladder, lymph node metastases are rare in non-muscle invasive disease. Information regarding indications, extent and possible curative potential is currently lacking for lymphadenectomy in conjunction with nephroureterectomy for urothelial carcinoma in the upper urinary tract (UUTUC). There are, however, retrospective series with survival data for patients with lymph node metastasis that report long term survival after surgery as monotherapy with similar survival proportions as in bladder cancer with lymph node metastases after radical cystectomy. A retrospective study from Tokyo was expanded to the only available prospective study, where 68 patients with UUTUC were submitted to template-based lymphadenectomy. Another retrospective study by the same Japanese group, showed that 5-year cancer-specific and recurrence-free survival was significantly higher in the complete lymphadenectomy group than in the incomplete lymphadenectomy or without lymphadenectomy groups. Tanaka N et al. reported recurrence rate after nephroureterectomy without lymphadenectomy at 1 and 3 years were 18.9 and 29.8 %, respectively.

Hypothesis: Complete lymphadenectomy during nephroureterectomy because of invasive urothelial carcinoma may reduce the incidence of lymph nodes metastasis, local recurrence, distant metastasis and improve the cancer survival rate.

Purpose: To evaluate the influence of complete lymphadenectomy on recurrence and cancer specific survival rate compared to limited or no lymphadenectomy.

Primary endpoint/analysis: Recurrence free survival at five-year postoperative. Secondary endpoints: Incidence of lymph node metastases, local recurrence and/or distant metastasis, cancer specific and overall survival at one, three and five-year postoperative. Complications rate according to Clavien classification within the first thirty days postoperatively.

Another endpoint/analysis: Multivariate analysis of possible preoperative risk factors for lymph node metastases (tumour size, preoperative urinary cytology, lymph node enlargement on CT, PET-CT positivity) and postoperative risk factors for lymph node metastases (stage, grade, tumour diameter, presence of necrosis in the tumour (none; <10%; >10% of total tumour area), number of lymph nodes excised).

Design: Prospectively randomized to template based lymphadenectomy or not, in patients with clinically muscle-invasive UUTUC in the renal pelvis or upper 2/3 of the ureter. One to one, controlled clinical trial. Patients will be randomly allocated into two groups, 183 patients in each group. Group A will be scheduled to receive routine standard open or robot assisted nephroureterectomy without lymphadenectomy except for clinically enlarged. Group B will be scheduled to received mapped lymphadenectomy in conjugation with nephroureterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Locally advanced high grade urothelial carcinoma in the renal pelvis or upper 2/3 of the ureter (Clinical stage > T1)
3. Patient with ECOG performance score of 2 and less.
4. Able to give informed consent

Exclusion Criteria:

1. Clinical suspicion of non-muscle invasive UUTUC
2. Metastatic urothelial carcinoma for the renal pelvis or upper 2/3 of the ureter
3. Inability to understand written consent forms or give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | Five years

SECONDARY OUTCOMES:
Incidence of metastasis | Five years

OTHER OUTCOMES:
Complications | Within 30 days after operations

CONTACTS AND LOCATIONS:
Overall Officials: Nessn H Azawi, MB.Ch.B., Study Chair — Roskilde University Hospital
Locations (1):
- Roskilde Hospital, Roskilde, Denmark

REFERENCES:
- [Background] Holmang S, Johansson SL. Bilateral metachronous ureteral and renal pelvic carcinomas: incidence, clinical presentation, histopathology, treatment and outcome. J Urol. 2006 Jan;175(1):69-72; discussion 72-3. doi: 10.1016/S0022-5347(05)00057-1. PMID 16406872
- [Background] Hall MC, Womack S, Sagalowsky AI, Carmody T, Erickstad MD, Roehrborn CG. Prognostic factors, recurrence, and survival in transitional cell carcinoma of the upper urinary tract: a 30-year experience in 252 patients. Urology. 1998 Oct;52(4):594-601. doi: 10.1016/s0090-4295(98)00295-7. PMID 9763077
- [Background] Olgac S, Mazumdar M, Dalbagni G, Reuter VE. Urothelial carcinoma of the renal pelvis: a clinicopathologic study of 130 cases. Am J Surg Pathol. 2004 Dec;28(12):1545-52. doi: 10.1097/00000478-200412000-00001. PMID 15577672
- [Background] Lughezzani G, Jeldres C, Isbarn H, Shariat SF, Sun M, Pharand D, Widmer H, Arjane P, Graefen M, Montorsi F, Perrotte P, Karakiewicz PI. A critical appraisal of the value of lymph node dissection at nephroureterectomy for upper tract urothelial carcinoma. Urology. 2010 Jan;75(1):118-24. doi: 10.1016/j.urology.2009.07.1296. Epub 2009 Oct 28. PMID 19864000
- [Background] Kondo T, Nakazawa H, Ito F, Hashimoto Y, Toma H, Tanabe K. Primary site and incidence of lymph node metastases in urothelial carcinoma of upper urinary tract. Urology. 2007 Feb;69(2):265-9. doi: 10.1016/j.urology.2006.10.014. PMID 17320661
- [Background] Kondo T, Hara I, Takagi T, Kodama Y, Hashimoto Y, Kobayashi H, Iizuka J, Omae K, Ikezawa E, Yoshida K, Tanabe K. Possible role of template-based lymphadenectomy in reducing the risk of regional node recurrence after nephroureterectomy in patients with renal pelvic cancer. Jpn J Clin Oncol. 2014 Dec;44(12):1233-8. doi: 10.1093/jjco/hyu151. Epub 2014 Sep 30. PMID 25271269
- [Background] Tanaka N, Kikuchi E, Kanao K, Matsumoto K, Kobayashi H, Ide H, Miyazaki Y, Obata J, Hoshino K, Shirotake S, Akita H, Kosaka T, Miyajima A, Momma T, Nakagawa K, Hasegawa S, Nakajima Y, Jinzaki M, Oya M. Metastatic behavior of upper tract urothelial carcinoma after radical nephroureterectomy: association with primary tumor location. Ann Surg Oncol. 2014 Mar;21(3):1038-45. doi: 10.1245/s10434-013-3349-z. Epub 2013 Nov 12. PMID 24217788
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542